CLINICAL TRIAL: NCT06564558
Title: The Effect of Postural Correctional Interventions on the Quality of Life of Patients With Gastroesophageal Reflux Disease.
Brief Title: The Effect of Postural Correction On Gastroesophageal Reflux Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Associate Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: GERD QoL
Record Dates: First submitted 2024-07-07; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Gastro Esophageal Reflux; Gastro Esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: The study will follow a randomized controlled clinical trial design. Participants will be recruited from the physical therapy outpatient clinic at Beirut Arab University as well as several outpatient and private physical therapy clinics around Beirut, Lebanon. After recruitment and screening for eligibility, the participants will be divided randomly using a computer randomization program into a control and experimental group. After the completion of the program, the two groups will be compared based on selected outcome measures.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Postural Correction Group (Experimental): The experimental group will receive real thoracic spine hyperkyphosis treatment. This treatment is focused around impairments that are linked with spinal kyphosis such as spinal extensor muscle weakness, anterior muscle chain tightness, and thoracic spine hypomobility. The participants will undergo spinal strengthening exercises, thoracic spine tight musculature stretching, and finally thoracic spine mobility exercises. All exercises will follow a 3 set parameter rule with patient tolerance kept in mind.
  Interventions: Other: Spinal Strengthening Exercises; Other: Thoracic Spine Stretching; Other: Thoracic Spine Mobilization
- Sham Postural Correction Group (Sham Comparator): The control group will receive sham thoracic kyphosis treatment comprised an hour of social interaction with similar participants where a blinded therapist will provide educational tips for dealing with kyphosis along with educational reading material for each participant.
  Interventions: Other: Sham Postural Correction

INTERVENTIONS:
Other: Spinal Strengthening Exercises — Individuals in the experimental group will carry out 3 sets of 10 repetitions or what is tolerated within a Borg scale intensity of 4-5 with 70-80% of perceived exertion with appropriately picked elastic bands. The exercises include: Shoulder horizontal abduction; Shoulder elevation; Back Extensions over a plinth; Shoulder extension exercises; One arm and opposite leg lifts from quadruped; and finally bilateral arm lifts with upper thoracic extension from prone (superman exercise).
  Arms: Real Postural Correction Group
Other: Thoracic Spine Stretching — Participants will be instructed to do two exercises: Firstly, to lay supine with and hinge the thoracic spine over a roller placed in a way that would ensure the patient is forward lying and not completely supine. The participant will be instructed to maintain hinging until a stretch or pressure feeling is felt in the midback and hold this position for 3 sets of 30 seconds. Secondly, the patient was asked to be in a seated position, clasp the hands together and behind the head while arching backward over the chair and looking up. This exercise will be done for 3 sets of 20-30 repetitions with a slight hold time at the end of the movement. All interventions will be carried out for 45 minute sessions 3 times per week.
  Arms: Real Postural Correction Group
Other: Thoracic Spine Mobilization — The patient will be seated with both hands clasped at shoulder level. An experienced and blinded therapist standing homolateral to the patient supports the clasped hands with one arm while placing the other hand was placed at different thoracic regions until the thoracolumbar junction. Specifically, the dorsal aspect of the index finger and pad of the thumb were used to create a fixation point at the junction. Following that, gentle extension-directed glides (postero-anterior) will be done by the therapist for 3 sets of 10 repetitions or until tolerated by the patient.
  Arms: Real Postural Correction Group
Other: Sham Postural Correction — comprised an hour of social interaction with similar participants where a blinded therapist will provide educational tips for dealing with kyphosis along with educational reading material for each participant.
  Arms: Sham Postural Correction Group

SUMMARY:
The main aim of this randomized controlled trial is to investigate the effects of postural correctional exercises and interventions on the severity of symptoms of gastroesophageal reflux disease (GERD) as well as the quality of life of patients afflicated with this disease. The main questions this study aims to answer is:

1. Do postural correctional exercises reduce the symptoms of GERD?
2. Do postural correctional exercises improve the quality of life of individuals afflicted with GERD?

The experimental group in this study will undergo real postural correctional exercises whereas the control group will undergo sham postural correctional interventions and then the two groups will be compared post-treatment based on GERD severity of symptoms as well as quality of life of the patients afflicted with GERD.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a disease that occurs when the normal physiological process termed gastroesophageal reflux (GER) begins to cause painful, harmful, or irritating signs and symptoms to certain individuals. This happens when the defence lines composed mainly of the lower esophageal sphincter (LES) and the angle of His are affected by a multitude of factors. These include abnormal resting pressure of the LES, increase intra-abdominal pressure compared to the resting pressure of the LES, certain medication side effects, and certain body positioning. The latter combined with posture has also been pointed out as a factor that might affect GERD by affecting the angle of His that acts similar to a valve between the esophagus and the curvature of the stomach.

Several works of literature have found a link between GERD and postural abnormalities or deformities. Scoliosis, defined as a spinal deformity consisting of a lateral curvature with or without rotation of the vertebra, has been shown to be a risk factor of GERD. More specifically, a left-sided thoracolumbar or lumbar lateral curvature, especially when greater than 30 degrees, has been cited by several studies as a risk factor for consideration with regards to GERD.

Accordingly, a certain relationship might be present between spinal deformities and/or abnormal spinal positioning, more specifically in the thoracic and thoracolumbar regions, and severity as well as prevalence of GERD. As such, the aim of this study is to investigate the effect of postural correctional interventions (PCI) on severity of GERD symptoms and quality of life in patients afflicted with the disease.

The experimental group in this study will undergo real postural correctional exercises whereas the control group will undergo sham postural correctional interventions and then the two groups will be compared post-treatment based on GERD severity of symptoms as well as quality of life of the patients afflicted with GERD.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 60.
* Diagnosed with GERD by a primary medical doctor.
* Patients with a kyphosis angle greater than 30 degrees.
* A score of 8 or greater on the Frequency Scale for the Symptoms of GERD (FSSG) which is considered positive.

Exclusion Criteria:

* Individuals with recent spinal surgery.
* Recent spinal trauma in the thoracic or lumbar regions
* A score less than 8 on the FSSG
* Having no associated thoracic or thoracolumbar deformity or abnormal alignment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Frequency Scale for the Symptoms of GERD (FSSG) | Taken initially before intervention process, at 6 months follow up and at 12 months follow up.
  The Frequency Scale for the Symptoms of GERD is a scale comprised of 12 questions targeted at assessing the severity of GERD symptoms. Each question is scored on an ordinal basis as follows: never=0; occasionally=1; sometimes=2; often=3; and always=4. The questions include statements such as: "do you get heartburn" and "do you get a bitter liquid (acid) coming up into your throat. This scale has been used widely in the literature that had similar aims to this study in assessing the severity of GERD.

SECONDARY OUTCOMES:
Kyphosis Cobb Angle Assessment Using X-ray Radiographs: | Taken initially before intervention process, at 6 months follow up and at 12 months follow up.
  Initially the Cobb angle was created to measure scoliosis, however with the adjustment of the patient position and plane of radiography it has been proven useful to assess kyphosis and hyperkyphosis. At this time, the Cobb angle assessed using X-ray radiographs is considered the golden standard for kyphosis assessment. The patient will be standing with the X-ray taken at the side by a licensed and experienced technician. The Cobb angle will then be computed and given to the outcome assessors.
GERD Quality of Life Questionnaire (GERD QOL) | Taken initially before intervention process, at 6 months follow up and at 12 months follow up.
  The GERD Quality of Life Questionnaire is a 16-item questionnaire encompassing 4 different areas daily activity, treatment effect, diet, and psychological well-being. Each are is scored on a scale of 0 to 4 meaning the following: 0= Strongly Agree, 1= Agree, 2= Neutral, 3= Disagree, 4= Strongly Disagree. The higher the score the lesser the impact of GERD on quality of life and thus the better score. After answering each question, all the questions corresponding to each aspect are summed and divided by the maximum score attainable and divided by 100. The total scores for each aspect are then added up and divided by 4 to get a final score. This questionnaire was proven to have good validity and reliability in assessing the impact of GERD on patient quality of life.
Short Forum Suvery SF-12v2: | Taken initially before intervention process, at 6 months follow up and at 12 months follow up.
  General health related quality of life will be assessed using the SF-12v2 questionnaire which is a simplified and shortened version of the SF-36 questionnaire. The questionnaire contains 12 questions over eight different health-related domains. Each of the 8 domains or subscales is scored from 0-100 with higher scores indicating better health. In addition to the 8 subscale scores, the SF12v2 is reportedly capable of reporting summary scores for physical and mental health individually with scores also ranging from 0-100 and higher scores indicating better health. The questionnaire was described as both valid and reliable in recent literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided